CLINICAL TRIAL: NCT03578666
Title: Effects of Massage and Cold Water Immersion After Exhausting Exercise on Biomechanical Parameters and Running Economy: A Randomized Controlled Trial
Brief Title: Massage Versus Cold Water Immersion for Fatigue-induced Biomechanical Alterations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iraia Bidaurrazaga-Letona (Other)
Responsible Party: Sponsor-Investigator, Iraia Bidaurrazaga-Letona, PhD, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IT811-13
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Running; Fatigue
Keywords: recovery intervention; fatigue; running; cryotherapy; running economy
MeSH Terms: conditions — Fatigue | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage Group (Experimental): Recreational active runners recruited from local running clubs (n= 16) will receive 40 minutes of massage therapy.
  Interventions: Other: Massage
- Cold water immersion group (Experimental): Recreational active runners recruited from local running clubs(n= 16) will immerse for 10 minutes in a cold water bath
  Interventions: Other: Cold water immersion
- Control group (No Intervention): Recreational active runners recruited from local running clubs will rest passively in a sitting position for 30-min period

INTERVENTIONS:
Other: Massage — The intervention will be applied to both legs to a constant distal to proximal stroking rhythm. Firstly, participants will be lying in a prone position for 22 min: 1 min on the sole of the foot, 1 min on the Achilles tendon, 1 min on the soleus muscle, 3 min on the triceps muscle, 4 min on the hamstring muscles, 30 s tapotement from the sole of the foot to the hamstrings and 30 s superficial effleurage from the sole of the foot to the hamstrings. Then they will assume a supine position for 18 min: 1 min on the sole of the foot, 3 min on the tibialis anterior and peroneus lateralis muscles and 4 min in the quadriceps, adductors and lata muscles, 30 s tapotement from the sole of the foot to the hamstrings and 30 s superficial effleurage from the sole of the foot to the hamstrings.
  Arms: Massage Group
Other: Cold water immersion — The cold water immersion group immersed their lower limbs (ensuring that the iliac crests were fully immersed) in an ice bath filled with cooled water for 10 min. The water was maintained at a mean temperature of 10 degrees (±0.5°) by the addition of ice.
  Arms: Cold water immersion group

SUMMARY:
The optimization of recovery to alleviate the effects of fatigue in athletes can provide valuable performance advantage. However, despite the growing body of literature regarding effects of different interventions in fatigue, there is still lack of clarity regarding the efficacy of interventions on running economy and, particularly, fatigue-induced biomechanical alterations. Therefore, the aim of this study was to compare the effects of massage and cold water immersion for enhancing recovery and alleviating fatigue after an exhausting training session. We hypothesized that both massage and cold water immersion would enhance biomechanical parameters compared with a control condition and hence would improve subsequent running economy.

DETAILED DESCRIPTION:
In this randomized controlled all the subjects (n=48) will performed the same protocol. The protocol will begin with a exhausting training session (20-min warm-up consisted of 15-min of continuous self-paced running followed by 5-min of fast-finish progression runs increasing speeds (from approximately 60% to 80% of maximal heart rate, participant controlled), 10 x 500 m sprints at 90% of maximal heart rate with a 2-min rest period between bouts and a recovery phase consisting of 10-min of slow jogging). Twenty-four hours after this exhausting training, subjects will perform an incremental running test on a treadmill (Pre-intervention test) where subjects will start at 12 km/h for 6 min after which speed will be increased by 2 km/h every 6 min until a 16 km/h trial is completed. At the end of each stage, participants will rate their perceived exertion using the 10-point Modified Borg rating of perceived exertion scale (RPE scale). One hour after this test, in one protocol subjects will receive the massage intervention, (Massage group); other group will receive a cold water immersion intervention (Cold water immersion group); in the other group (Control group) participants will rest passively in a sitting position for 30-min period. To evaluate the relevance of the changes induced by the interventions (massage, cold water immersion, passive rest) subjects will repeat the treadmill test 48 hours after the first test (72 hours after the exhaustive training).

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (current participation in races and a 10-km race time<34.5-min)

Exclusion Criteria:

* Suffered from any injury within the preceding 4 months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
- CHANGE FROM BASELINE OXYGEN UPTAKE AT 48 HOURS AFTER THE TREATMENT | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Oxygen uptake (mL kg-1 min-1) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Oxygen uptake will be recorded using a gas analyzer system (Esgostik Geratherm, Geschwenda, Germany).
- CHANGE FROM BASELINE STRIDE LENGTH AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride length (cm) defined as the length the treadmill belt moves from toe-off to initial ground contact in successive steps, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE STRIDE FREQUENCY AT 48 HOURS AFTER THE TREATMENT. | Time Frame: Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride frequency, defined as the number of ground contact events per minute, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE STRIDE ANGLE AT 48 HOURS AFTER THE TREATMENT. | Time Frame: Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride angle (º), defined as the angle of the parable tangent derived from the theoretical arc traced by a foot during a stride and the ground, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE GROUND CONTACT TIME AT 48 HOURS AFTER THE TREATMENT. | Time Frame: Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Ground contact time (s), defined as the time from when the foot contacts the ground to when the toes left the ground and was determined by the disruption of the infrared gates, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE SWING TIME AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  The swing time (ms) corresponds to the time from foot flat to initial take-off. Swing time will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE CONTACT PHASE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Contact time (ms), defined as the percentage of the ground contact time at which the different sub-phases of stance phase occur, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
- CHANGE FROM BASELINE RATING OF PERCEIVED EXERTION AT 48 HOURS AFTER THE TREATMENT | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Modified Borg rating of perceived exertion scale (RPE scale) defined as a way of measuring physical activity intensity level, how hard you feel like your body is working. The Borg RPE scale is a numerical scale that ranges from 1 to 10, where 0 means "no exertion at all" and 10 means "maximal exertion."

SECONDARY OUTCOMES:
Body height (cm) | Participants will be assessed at baseline (24 hours after an exhaustive training session).
  - Body height (cm) will be measured using a stadiometer (Año Sayol, Barcelona, Spain) following the guidelines outlined by the International Society for the Advancement of Kinanthropometry.
Body mass (kg) | Participants will be assessed at baseline (24 hours after an exhaustive training session).
  - Body mass (kg) will be measured using a balance (Año Sayol, Barcelona, Spain) following the guidelines outlined by the International Society for the Advancement of Kinanthropometry.
- Skinfolds (mm) | Participants will be assessed at baseline (24 hours after an exhaustive training session).
  - Skinfolds (mm) will be measured at four sites (triceps, subscapular, abdominal, suprailiac) using a Harpenden Skinfold Caliper (Baty, West Sussex, UK) following the guidelines outlined by the International Society for the Advancement of Kinanthropometry.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunabeitia I, Arrieta H, Rodriguez-Larrad A, Gil J, Esain I, Gil SM, Irazusta J, Bidaurrazaga-Letona I. Effects of Massage and Cold Water Immersion After an Exhaustive Run on Running Economy and Biomechanics: A Randomized Controlled Trial. J Strength Cond Res. 2022 Jan 1;36(1):149-155. doi: 10.1519/JSC.0000000000003395. PMID 31800477